CLINICAL TRIAL: NCT00822120
Title: A Phase II Trial of Response-Adapted Therapy of Stage III-IV Hodgkin Lymphoma Using Early Interim FDG-PET Imaging
Brief Title: S0816 Fludeoxyglucose F 18-PET/CT Imaging and Combination Chemotherapy With or Without Additional Chemotherapy and G-CSF in Treating Patients With Stage III or Stage IV Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000630501; S0816 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Lymphoma; Nonneoplastic Condition
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; HIV infection
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; HIV Infections | interventions — Bleomycin; Filgrastim; ABVD protocol; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Prednisone; Procarbazine; Vinblastine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HIV Positive, PET Positive: BEACOPP standard (Experimental): Etoposide 100 mg/m2 IV Days 1, 2, 3 Dox 25 mg/m2 IV Day 1 Cyclo 650mg/m2 IV Day 1 Procarb 100 mg/m2 PO Days 1-7 Pred 40 mg/m2 PO Days 1-14 Bleo 10u/m2 IV Day 8 Vincristine 1.4 mg/m2 IV Day 8 Q 21 Days x 6 cycles
  Interventions: Biological: bleomycin sulfate; Drug: BEACOPP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate
- HIV Negative, PET Positive: BEACOPP escalated (Experimental): Etoposide 200 mg/m2 IV Days 1, 2, 3 Dox 35 mg/m2 IV Day 1 Cyclo 1,250 mg/m2 IV Day 1 Procarb 100 mg/m2 PO Days 1-7 Pred 40 mg/m2 PO Days 1-14 Bleo 10u/m2 IV Day 8 Vincristine 1.4 mg/m2 IV Day 8 G-CSF 5mcg/kg/day SQ Days 8-14 Q 21 Days x 6 cycles
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: BEACOPP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate
- HIV Positive, PET Negative: ABVD (Active Comparator): Doxorubicin 25 mg/m2 IV Bleomycin 10u/m2 IV Vinblastine 6mg/m2 IV Dacarbazine 375 mg/m2 IV Days 1, 15 Q 28 Days x 2
  Interventions: Biological: bleomycin sulfate; Drug: ABVD regimen; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine sulfate
- HIV Negative, PET Negative: ABVD (Active Comparator): Doxorubicin 25 mg/m2 IV Bleomycin 10u/m2 IV Vinblastine 6mg/m2 IV Dacarbazine 375 mg/m2 IV Days 1, 15 Q 28 Days x 2
  Interventions: Biological: bleomycin sulfate; Drug: ABVD regimen; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine sulfate

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
  Arms: HIV Negative, PET Positive: BEACOPP escalated
Drug: ABVD regimen
  Arms: HIV Negative, PET Negative: ABVD; HIV Positive, PET Negative: ABVD
Drug: BEACOPP regimen
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard
Drug: cyclophosphamide
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard
Drug: dacarbazine
  Arms: HIV Negative, PET Negative: ABVD; HIV Positive, PET Negative: ABVD
Drug: doxorubicin hydrochloride
Drug: etoposide
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard
Drug: prednisone
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard
Drug: procarbazine hydrochloride
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard
Drug: vinblastine sulfate
  Arms: HIV Negative, PET Negative: ABVD; HIV Positive, PET Negative: ABVD
Drug: vincristine sulfate
  Arms: HIV Negative, PET Positive: BEACOPP escalated; HIV Positive, PET Positive: BEACOPP standard

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. G-CSF may help lessen the side effects in patients receiving chemotherapy. Imaging procedures, such as fludeoxyglucose F 18-PET/CT imaging, may help doctors predict how patients will respond to treatment.

PURPOSE: This phase II trial is studying fludeoxyglucose F 18-PET/CT imaging to see how well it works in assessing response to combination chemotherapy and allow doctors to plan better additional further treatment in treating patients with stage III or stage IV Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the 2-year progression-free survival (PFS) of HIV-negative patients with stage III-IV Hodgkin lymphoma treated with response-adapted therapy based on fludeoxyglucose F 18 (FDG)-PET imaging after 2 courses of doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine (ABVD).
* To estimate the 2-year PFS of patients who are PET-positive after treatment with 2 courses of ABVD and an escalated dose regimen comprising cyclophosphamide, doxorubicin hydrochloride, etoposide, vincristine sulfate, bleomycin, procarbazine hydrochloride, and prednisone (BEACOPP).

Secondary

* To estimate the 2-year overall survival (OS) of patients treated with these regimens.
* To estimate the response rate (i.e., complete and partial responses) in patients treated with these regimens.
* To evaluate the toxicity of these response-adapted regimens.
* To document the feasibility of centralized, real-time review of FDG-PET imaging for U.S. cooperative group studies.
* To prospectively evaluate the overall response rate, complete response rate, PFS, and OS of HIV-positive patients treated with these response-adapted regimens.

OUTLINE: This is a multicenter study.

All patients undergo baseline whole-body fludeoxyglucose F 18 (FDG)-PET/CT imaging before beginning chemotherapy. Patients then receive doxorubicin hydrochloride IV, bleomycin IV, vinblastine IV, and dacarbazine IV (ABVD) on days 1 and 15. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Between days 22 and 25 of course 2, patients undergo a second FDG-PET/CT scan to assess response. Subsequent therapy is based on FDG-PET/CT scan results. Patients are stratified according to FDG-PET positivity (yes vs no). Patients who are FDG-PET-negative continue treatment with ABVD for up to 4 additional courses in the absence of disease progression or unacceptable toxicity. Patients who are FDG-PET-positive are then further stratified according to HIV positivity (yes or no) and receive 1 of the following treatment regimens:

* Escalated-dose BEACOPP chemotherapy: HIV-negative patients receive escalated-dose BEACOPP chemotherapy comprising doxorubicin hydrochloride IV and cyclophosphamide IV on day 1, etoposide IV on days 1-3, oral procarbazine hydrochloride on days 1-7, oral prednisone on days 1-14, and bleomycin IV and vincristine IV on day 8. Patients receive filgrastim (G-CSF) subcutaneously on days 8-14. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Standard-dose BEACOPP chemotherapy: HIV-positive patients receive standard dose BEACOPP chemotherapy comprising doxorubicin hydrochloride IV and cyclophosphamide IV on day 1, etoposide IV on days 1-3, oral procarbazine hydrochloride on days 1-7, oral prednisone on days 1-14, and bleomycin IV and vincristine IV on day 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Six to eight weeks after completion of chemotherapy, patients undergo a post-treatment FDG-PET/CT scan.

Some patients may undergo bone marrow biopsy at 1 month after the last course of chemotherapy.

After completion of study treatment, patients are followed up periodically for 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin lymphoma (HL) (i.e., nodular sclerosis, mixed cellularity, lymphocyte-rich, or lymphocyte-depleted)

  * Previously untreated stage III or IV disease
  * No nodular lymphocyte predominant disease
* Bidimensionally measurable disease
* Adequate biopsy samples from original diagnostic specimen must be available for pathologic review

  * Tissue obtained from core biopsies allowed
  * No tissue obtained from needle aspirations or cytologies
* Must have known HIV status

  * No multi-drug resistant HIV infection, CD4 counts < 150/μL, or other concurrent AIDS-defining conditions in HIV-positive patients
  * HIV-positive patients with CD4 counts ≥ 150/μL at the time of enrollment OR documented CD4 count > 250/μL at any time within 8 months prior to HL diagnosis allowed
* Must have undergone unilateral or bilateral bone marrow biopsy within the past 42 days
* Must have a diagnostic quality CT scan of the chest/abdomen and pelvis AND baseline FDG-PET scan within the past 28 days

  * Combined PET/CT scans required
  * No older "stand-alone" FDG-PET scans
  * No low-resolution "localization" CT scans as part of a combined PET/CT scans

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Serum erythrocyte sedimentation rate, lactate dehydrogenase (LDH), hemoglobin, albumin, white blood cell count (WBC), and lymphocytes measured within the past 28 days
* Serum estradiol (women only), testosterone (men only), follicle stimulating hormone (FSH) and luteinizing hormone (LH) (both men and women) levels must be drawn within 60 days prior to registration
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* No significant cardiac abnormalities as assessed by multiple gated acquisition scan (MUGA) or ECHO AND cardiac ejection fraction ≥ 45% in patients with a history of hypertension or cardiac symptoms
* Hepatitis B-negative (i.e., hepatitis B surface antigen-negative or anti-hepatitis B core antigen-negative)

  * Patients immune to or immunized against hepatitis B (i.e., anti-hepatitis B surface antibody-positive) are eligible
* Hepatitis C-negative (i.e., anti-hepatitis C antibody-negative)
* No significant lung disease with abnormal lung function tests (i.e., diffusing capacity of lung for carbon monoxide (DLCO) > 25% below predicted after correction for hemoglobin) unless attributable to lymphoma
* No requirement for continuous supplemental oxygen therapy
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, radiotherapy, or antibody therapy for lymphoma
* No prior solid organ transplantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 371 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W. Press, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (423):
- United States (423):
  - Arizona Cancer Center at University Medical Center North, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Springdale, Rogers, Arkansas
  - Kaiser Permanente Medical Center - Anaheim/Orange County, Anaheim, California
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Kaiser Permanente Medical Center - Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Medical Center - Fontana, Fontana, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Kaiser Permanente Medical Center - Harbor City, Harbor City, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Kaiser Permanente - Irvine, Irvine, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Kaiser Foundation Hospital - West Los Angeles, Los Angeles, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Group, Panorama City, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Riverside, Riverside, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Kaiser Permanente Medical Cener - Woodland Hills, Woodland Hills, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Regional Medical Center, Lewiston, Idaho
  - Idaho Urologic Institute, PA, Meridian, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Delnor Hospital - Geneva, Geneva, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Central Dupage Cancer Center, Warrenville, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Ministry Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Stephens DM, Li H, Schoder H, Straus DJ, Moskowitz CH, LeBlanc M, Rimsza LM, Bartlett NL, Evens AM, LaCasce AS, Barr PM, Knopp MV, Hsi ED, Leonard JP, Kahl BS, Smith SM, Friedberg JW. Five-year follow-up of SWOG S0816: limitations and values of a PET-adapted approach with stage III/IV Hodgkin lymphoma. Blood. 2019 Oct 10;134(15):1238-1246. doi: 10.1182/blood.2019000719. PMID 31331918
- [Derived] Hsi ED, Li H, Nixon AB, Schoder H, Bartlett NL, LeBlanc M, Smith S, Kahl BS, Leonard JP, Evens AM, Scott DW, Rimsza LM, Friedberg JW. Serum levels of TARC, MDC, IL-10, and soluble CD163 in Hodgkin lymphoma: a SWOG S0816 correlative study. Blood. 2019 Apr 18;133(16):1762-1765. doi: 10.1182/blood-2018-08-870915. Epub 2019 Feb 5. PMID 30723079

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-negative: Initial ABVD; HIV-positive: Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles
- HIV-negative and PET-negative: Continued ABVD; HIV-positive and PET-negative: Continued ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles
- HIV-negative and PET-positive: BEACOPP Escalated: Etoposide 200 mg/m^2 IV Days 1, 2, 3, Doxorubicin 35 mg/m^2 IV Day 1, Cyclophosphamide 1,250 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, G-CSF 5mcg/kg/day SQ Days 8-14, Q 21 Days x 6 cycles
- HIV-positive and PET-positive: BEACOPP Standard: Etoposide 100 mg/m^2 IV Days 1, 2, 3, Doxorubicin 25 mg/m^2 IV Day 1, Cyclophosphamide 650 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, Q 21 Days x 6 cycles
Period: Initial Registration
Arm/Group | HIV-negative: Initial ABVD | HIV-positive: Initial ABVD | HIV-negative and PET-negative: Continued ABVD | HIV-negative and PET-positive: BEACOPP Escalated | HIV-positive and PET-negative: Continued ABVD | HIV-positive and PET-positive: BEACOPP Standard
Started | 358 | 13 | 0 | 0 | 0 | 0
Eligible and Evaluable Patients | 336 | 12 | 0 | 0 | 0 | 0
Completed | 332 | 12 | 0 | 0 | 0 | 0
Not Completed | 26 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal Unrelated to Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Reasons not Protocol Specified | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 22 | 1 | 0 | 0 | 0 | 0
Period: PET-directed Therapy
Arm/Group | HIV-negative: Initial ABVD | HIV-positive: Initial ABVD | HIV-negative and PET-negative: Continued ABVD | HIV-negative and PET-positive: BEACOPP Escalated | HIV-positive and PET-negative: Continued ABVD | HIV-positive and PET-positive: BEACOPP Standard
Started | 0 | 0 | 270 | 55 | 10 | 1
Eligibile and Evaluable Patients | 0 | 0 | 270 | 55 | 10 | 1
Completed | 0 | 0 | 270 | 45 | 10 | 1
Not Completed | 0 | 0 | 0 | 10 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Refusal Unrelated to Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible and evaluable HIV-positive patients were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV-negative: Initial ABVD | HIV-positive: Initial ABVD | Total
Number analyzed (Participants) | 336 | 12 | 348
Age, Continuous [Median (Full Range); unit: years] | 32.1 [18 to 60] | 44.6 [25 to 50] | 32.4 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 2 | 149
  Male | 189 | 10 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 3 | 31
  Not Hispanic or Latino | 273 | 8 | 281
  Unknown or Not Reported | 35 | 1 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 32 | 4 | 36
  White | 274 | 5 | 279
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HIV-negative Patients With 2-year Progression-free Survival (PFS) Treated With 2 Initial Cycles of Adriamycin, Bleomycin, Vnblastine, and Dacarbazine (ABVD) Followed by Response-adapted Therapy Based on Interim FDG-PET Imaging.
Description: Disease progression is defined using the 2007 revised Cheson et al. criteria that is at least 50% increase in sum of the product of the diameters (SPD) of target measurable nodal lesions over the smallest sum observed, or >= 50% increase in greatest transverse diameter (GTD) of any nodal > 1 cm in shortest axis, or >= 50% increase in the SPD of other target measurable lesions over the smallest sum observed, any new bone marrow involvement, any new lesion, lymph node with long axis is > 1.5 cm or if both long and short axes are > 1 cm, PET positive if patients with no pretreatment PET scan or when PET scan was positive before therapy. Progression-free survival is measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 2 years
Population: Eligible and evaluable HIV-negative patients who started initial ABVD were included in the analysis regardless the response-adapted therapy after 2 initial cycles of ABVD was administered.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HIV-negative: 2 Cycles of ABVD Followed by PET-directed Therap: HIV-negative patients treated with 2 cycles of ABVD followed by response-adapted therapy. Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles. Interim PET-negative patients continue with 4 cycles of ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles. Interim PET-positive patients receive 6 cycles of escalated BEACOPP: Etoposide 200 mg/m^2 IV Days 1, 2, 3, Doxorubicin 35 mg/m^2 IV Day 1, Cyclophosphamide 1,250 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, G-CSF 5mcg/kg/day SQ Days 8-14, Q 21 Days x 6 cycles.
Arm/Group | HIV-negative: 2 Cycles of ABVD Followed by PET-directed Therap
Number analyzed (Participants) | 336
percentage of participants | 79 [74 to 83]

2. Primary Outcome: Percentage of HIV-negative Patients Who Are PET-positive After 2 Cycles of ABVD With 2-year PFS
Description: as for outcome 1
Time Frame: 2 years
Population: Eligible and evaluable HIV-negative patients who were PET-positive after 2 cycles of ABVD were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HIV-negative: 2 Cycles of ABVD Followed by Escalated BEACOPP: HIV-negative patients who are PET-positive are treated with 2 cycles of ABVD followed by escalated BEACOPP. Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles. Interim PET-positive patients receive 6 cycles of escalated BEACOPP: Etoposide 200 mg/m^2 IV Days 1, 2, 3, Doxorubicin 35 mg/m^2 IV Day 1, Cyclophosphamide 1,250 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, G-CSF 5mcg/kg/day SQ Days 8-14, Q 21 Days x 6 cycles.
Arm/Group | HIV-negative: 2 Cycles of ABVD Followed by Escalated BEACOPP
Number analyzed (Participants) | 60
percentage of participants | 64 [50 to 75]

3. Secondary Outcome: Percentage of HIV-negative Patients With 2-year Overall Survival (OS) Treated With 2 Initial Cycles of ABVD Followed by Response-Adapted Therapy Based on Interim FDG-PET Imaging
Description: Measured from date of registration to date of death due to any cause. Patients last known to be alive and are censored at date of last contact.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HIV-negative:2 Cycles of ABVD Followed by PET-directed Therapy: HIV-negative patients treated with 2 cycles of ABVD followed by response-adapted therapy. Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles. Interim PET-negative patients continue with 4 cycles of ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles. Interim PET-positive patients receive 6 cycles of escalated BEACOPP: Etoposide 200 mg/m^2 IV Days 1, 2, 3, Doxorubicin 35 mg/m^2 IV Day 1, Cyclophosphamide 1,250 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, G-CSF 5mcg/kg/day SQ Days 8-14, Q 21 Days x 6 cycles.
Arm/Group | HIV-negative:2 Cycles of ABVD Followed by PET-directed Therapy
Number analyzed (Participants) | 336
percentage of participants | 98 [95 to 99]

4. Secondary Outcome: Complete and Partial Response Rates for HIV-negative Patients Treated With Response- Adapted Therapy Based on FDG-PET Imaging After 2 Cycles of ABVD
Description: Complete Response (CR) is a complete disappearance of all disease with the exception of the following. If no PET scan or when the PET scan was positive before therapy, a post-treatment residual mass of any size is permitted if it is PET negative. If the PET scan was negative before therapy, all nodal masses at baseline must have regressed. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. Partial Response (PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes. If PET scan or when the PET scan was positive before therapy, PET should be positive in at least one previously involved site.
Time Frame: 7 months after registration
Population: Only eligible and evaluable HIV-negative patients who treated with response-adapted therapy based on FDG-PET imaging after 2 cycles of ABVD were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- PET-negative: Continued ABVD After 2 Cycles of ABVD: Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles Continued ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles
- PET-positive: BEACOPP Escalated After 2 Cycles of ABVD: Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles escalated BEACOPP: Etoposide 200 mg/m^2 IV Days 1, 2, 3, Doxorubicin 35 mg/m^2 IV Day 1, Cyclophosphamide 1,250 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, G-CSF 5mcg/kg/day SQ Days 8-14, Q 21 Days x 6 cycles
Arm/Group | PET-negative: Continued ABVD After 2 Cycles of ABVD | PET-positive: BEACOPP Escalated After 2 Cycles of ABVD
Number analyzed (Participants) | 270 | 55
percentage of patients | 100 [98.6 to 100] | 93 [82.4 to 97.9]

5. Secondary Outcome: Number of HIV-negative Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Up to 1 year
Population: Eligible HIV-negative patients who had received any treatment were included in the adverse event summaries. Six interim PET-positive patients who did not receive BEACOPP were excluded. patients Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-negative: Initial ABVD | HIV-negative and PET-negative: Continued ABVD | HIV-negative and PET-positive: BEACOPP Escalated
Number analyzed (Participants) | 336 | 270 | 49
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 3 | 0 | 0
  AST, SGOT | 1 | 0 | 0
  Adult respiratory distress syndrome (ARDS) | 0 | 2 | 0
  Albumin, serum-low (hypoalbuminemia) | 1 | 0 | 0
  Alkaline phosphatase | 1 | 0 | 0
  Allergic reaction/hypersensitivity | 2 | 2 | 0
  Anorexia | 1 | 1 | 0
  Arthritis (non-septic) | 1 | 0 | 0
  Carbon monoxide diffusion capacity (DL(co)) | 0 | 2 | 0
  Colitis | 0 | 1 | 0
  Colitis, infectious (e.g., Clostridium difficile) | 1 | 0 | 1
  Constipation | 1 | 0 | 0
  Cough | 0 | 1 | 0
  Creatinine | 0 | 0 | 1
  Cytokine release syndrome/acute infusion reaction | 1 | 0 | 0
  Dehydration | 1 | 2 | 1
  Diarrhea | 0 | 1 | 0
  Dizziness | 1 | 0 | 1
  Dyspnea (shortness of breath) | 4 | 9 | 1
  FEV(1) | 0 | 1 | 0
  Fatigue (asthenia, lethargy, malaise) | 10 | 15 | 3
  Febrile neutropenia | 8 | 17 | 17
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 0 | 3 | 1
  Glucose, serum-high (hyperglycemia) | 0 | 1 | 1
  Heartburn/dyspepsia | 1 | 0 | 0
  Hemoglobin | 10 | 4 | 37
  Hemolysis | 0 | 0 | 1
  Hemorrhage, pulmonary/upper respiratory - Nose | 0 | 0 | 1
  Hypotension | 0 | 0 | 1
  Hypoxia | 0 | 3 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 2 | 1 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 0 | 0 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 0 | 4 | 2
  Inf (clin/microbio) w/Gr 3-4 neuts - Meninges | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Mucosa | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 0 | 1 | 3
  Inf (clin/microbio) w/Gr 3-4 neuts - Soft tissue | 0 | 1 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - UTI | 0 | 1 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway | 0 | 1 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Vagina | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Catheter | 1 | 0 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 1 | 3 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - Oral cav | 0 | 0 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Skin | 1 | 0 | 1
  Infection with normal ANC or Grade 1 or 2 neutroph | 1 | 0 | 0
  Infection with unknown ANC - Lung (pneumonia) | 0 | 1 | 0
  Left ventricular systolic dysfunction | 0 | 1 | 0
  Leukocytes (total WBC) | 73 | 86 | 42
  Lymphopenia | 15 | 30 | 32
  Metabolic/Laboratory-Other (Specify) | 1 | 0 | 0
  Mood alteration - agitation | 1 | 0 | 0
  Mood alteration - anxiety | 1 | 0 | 0
  Mood alteration - depression | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1 | 0 | 2
  Mucositis/stomatitis (functional/symp) - Oral cav | 1 | 0 | 1
  Muscle weakness, not d/t neuropathy - body/general | 0 | 0 | 1
  Musculoskeletal/Soft Tissue-Other (Specify) | 0 | 1 | 0
  Nausea | 7 | 5 | 2
  Neuropathy: motor | 2 | 3 | 0
  Neuropathy: sensory | 4 | 12 | 4
  Neutrophils/granulocytes (ANC/AGC) | 206 | 165 | 38
  Osteonecrosis (avascular necrosis) | 0 | 0 | 1
  Pain - Abdomen NOS | 2 | 5 | 1
  Pain - Back | 1 | 0 | 3
  Pain - Bone | 0 | 0 | 5
  Pain - Cardiac/heart | 0 | 1 | 0
  Pain - Chest wall | 1 | 1 | 0
  Pain - Chest/thorax NOS | 0 | 1 | 1
  Pain - Extremity-limb | 1 | 0 | 0
  Pain - Head/headache | 2 | 2 | 0
  Pain - Joint | 1 | 0 | 1
  Pain - Muscle | 1 | 1 | 0
  Pain - Oral cavity | 1 | 0 | 0
  Pain - Skin | 0 | 1 | 0
  Pain - Stomach | 0 | 1 | 0
  Pain - Throat/pharynx/larynx | 0 | 0 | 1
  Pain - Tumor pain | 1 | 0 | 0
  Pain-Other (Specify) | 1 | 2 | 0
  Pancreatic endocrine: glucose intolerance | 1 | 1 | 0
  Phosphate, serum-low (hypophosphatemia) | 1 | 0 | 0
  Platelets | 1 | 0 | 34
  Pneumonitis/pulmonary infiltrates | 1 | 4 | 1
  Potassium, serum-high (hyperkalemia) | 0 | 0 | 1
  Potassium, serum-low (hypokalemia) | 0 | 0 | 4
  Rash/desquamation | 1 | 0 | 0
  Rigors/chills | 1 | 0 | 2
  Sodium, serum-low (hyponatremia) | 1 | 0 | 1
  Syncope (fainting) | 1 | 0 | 1
  Thrombosis/thrombus/embolism | 2 | 5 | 0
  Vomiting | 5 | 4 | 0
  Weight gain | 0 | 2 | 0

6. Secondary Outcome: Percentage of HIV-positive Patients With 2-year Progression-free Survival (PFS) Treated With Initial 2 Cycles of Adriamycin, Bleomycin, Vnblastine, and Dacarbazine (ABVD) Followed by Response-adapted Therapy Based on Interim FDG-PET Imaging.
Description: Disease progression is defined using the 2007 revised Cheson et al. criteria that is at least 50% increase in sum of the product of the diameters (SPD) of target measurable nodal lesions over the smallest sum observed, or >= 50% increase in greatest transverse diameter (GTD) of any nodal > 1 cm in shortest axis, or >= 50% increase in the SPD of other target measurable lesions over the smallest sum observed, any new bone marrow involvement, any new lesion, lymph node with long axis is >1.5 cm or if both long and short axes are > 1 cm, PET positive if patients with no pretreatment PET scan or when PET scan was positive before therapy. progression-free survival is measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 2 years
Population: Eligible and evaluable HIV-positive patients who started the initial ABVD were included in the analysis regardless the response-adapted therapy after 2 initial cycles of ABVD was administered.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- HIV-positive: 2 Cycles of ABVD Followed by PET-directed Therap: HIV-positive patients treated with 2 cycles of ABVD followed by response-adapted therapy. Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles. Interim PET-negative patients continue with 4 cycles of ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles. Interim PET-positive patients receive 6 cycles of standard BEACOPP: Etoposide 100 mg/m^2 IV Days 1, 2, 3, Doxorubicin 25 mg/m^2 IV Day 1, Cyclophosphamide 650 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, Q 21 Days x 6 cycles
Arm/Group | HIV-positive: 2 Cycles of ABVD Followed by PET-directed Therap
Number analyzed (Participants) | 12
percentage of patients | 83 [46 to 95]

7. Secondary Outcome: Percentage of HIV-positive Patients With 5-year Overall Survival (OS) Treated With 2 Initial Cycles of ABVD Followed by Response-Adapted Therapy Based on Interim FDG-PET Imaging.
Description: as for outcome 3
Time Frame: 5 years
Population: Eligible and evaluable HIV-positive patients who started initial ABVD were included in the analysis regardless the response-adapted therapy after 2 initial cycles of ABVD was administered.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HIV-positive: 2 Cycles of ABVD Followed by PET-directed Therap
Number analyzed (Participants) | 12
percentage of participants | 89 [43 to 98]

8. Secondary Outcome: Complete and Partial Response Rates for HIV-positive Patients Treated With Response-Adapted Therapy Based on FDG-PET Imaging After 2 Cycles of ABVD
Description: as for outcome 4
Time Frame: 7 months after registration
Population: Eligible and evaluable HIV-positive patients who treated with 2 initial cycles of ABVD followed by response-adapted therapy based on interim FDG-PET imaging were included he analysis.
Measure: Count of Participants; unit: Participants
Groups:
- PET-positive: BEACOPP Standard After 2 Cycles of ABVD: Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles standard BEACOPP: Etoposide 100 mg/m^2 IV Days 1, 2, 3, Doxorubicin 25 mg/m^2 IV Day 1, Cyclophosphamide 650 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, Q 21 Days x 6 cycles
Arm/Group | PET-negative: Continued ABVD After 2 Cycles of ABVD | PET-positive: BEACOPP Standard After 2 Cycles of ABVD
Number analyzed (Participants) | 10 | 1
Participants
  Complete Response | 9 | 0
  Partial Response | 1 | 1

9. Secondary Outcome: Number of HIV-positive Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: as for outcome 5
Time Frame: Up to 1 year
Population: Eligible HIV-positive patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Initial ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 2 cycles
- PET-negative: Continued ABVD: Doxorubicin 25 mg/m^2 IV, Bleomycin 10u/m^2 IV, Vinblastine 6mg/m^2 IV, Dacarbazine 375 mg/m^2 IV Days 1,15 Q 28 Days x 4 cycles
- PET-positive: BEACOPP Standard: Etoposide 100 mg/m^2 IV Days 1, 2, 3, Doxorubicin 25 mg/m^2 IV Day 1, Cyclophosphamide 650 mg/m^2 IV Day 1, Procarbzine 100 mg/m^2 PO Days 1-7, Prednisone 40 mg/m^2 PO Days 1-14, Bleomycin 10u/m^2 IV Day 8, Vincristine 1.4 mg/m^2 IV Day 8, Q 21 Days x 6 cycles
Arm/Group | Initial ABVD | PET-negative: Continued ABVD | PET-positive: BEACOPP Standard
Number analyzed (Participants) | 12 | 10 | 1
Participants
  Anorexia | 0 | 1 | 0
  Dizziness | 0 | 1 | 0
  Fatigue (asthenia, lethargy, malaise) | 1 | 1 | 0
  Febrile neutropenia | 3 | 3 | 0
  Hemoglobin | 1 | 3 | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Eye NOS | 1 | 0 | 0
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 0 | 1 | 0
  Infection with unknown ANC - Urinary tract NOS | 0 | 0 | 1
  Insomnia | 1 | 0 | 0
  Leukocytes (total WBC) | 7 | 6 | 1
  Lymphopenia | 1 | 2 | 1
  Mood alteration - agitation | 1 | 0 | 0
  Mood alteration - anxiety | 1 | 0 | 0
  Muscle weakness, not d/t neuropathy - body/general | 1 | 0 | 0
  Neuropathy: motor | 0 | 1 | 0
  Neuropathy: sensory | 1 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 8 | 7 | 1
  Pain - Bone | 1 | 0 | 0
  Pain - Joint | 1 | 1 | 0
  Phosphate, serum-low (hypophosphatemia) | 1 | 1 | 0
  Platelets | 0 | 1 | 0
  Sodium, serum-low (hyponatremia) | 1 | 0 | 0
  Thrombosis/thrombus/embolism | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | HIV-negative: Initial ABVD | HIV-negative and PET-negative: Continued ABVD | HIV-negative and PET-positive: BEACOPP Escalated | HIV-positive: Initial ABVD | HIV-positive and PET-negative: Continued ABVD | HIV-positive and PET-positive: BEACOPP Standard
Serious Adverse Events (participants affected / at risk) | 1/336 | 6/270 | 2/49 | 1/12 | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 335/336 | 268/270 | 49/49 | 12/12 | 9/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-negative: Initial ABVD (N=336) | HIV-negative and PET-negative: Continued ABVD (N=270) | HIV-negative and PET-positive: BEACOPP Escalated (N=49) | HIV-positive: Initial ABVD (N=12) | HIV-positive and PET-negative: Continued ABVD (N=10) | HIV-positive and PET-positive: BEACOPP Standard (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood alteration - agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-negative: Initial ABVD (N=336) | HIV-negative and PET-negative: Continued ABVD (N=270) | HIV-negative and PET-positive: BEACOPP Escalated (N=49) | HIV-positive: Initial ABVD (N=12) | HIV-positive and PET-negative: Continued ABVD (N=10) | HIV-positive and PET-positive: BEACOPP Standard (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 17 | 16 | 3 | 3 | 0
Hemoglobin (Blood and lymphatic system disorders) | 171 | 161 | 44 | 6 | 7 | 1
Palpitations (Cardiac disorders) | 2 | 4 | 3 | 0 | 0 | 0
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 7 | 9 | 3 | 1 | 1 | 0
Ocular/Visual-Other (Eye disorders) | 10 | 15 | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 114 | 73 | 10 | 5 | 2 | 0
Dental: teeth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 34 | 40 | 15 | 3 | 5 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 4 | 3 | 0 | 0 | 0
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 4 | 1 | 0 | 1 | 0 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 28 | 30 | 5 | 0 | 1 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 36 | 25 | 13 | 2 | 1 | 1
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 27 | 12 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 203 | 173 | 29 | 4 | 6 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 32 | 28 | 4 | 1 | 1 | 0
Pain - Oral cavity (Gastrointestinal disorders) | 14 | 4 | 5 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 68 | 74 | 19 | 3 | 4 | 0
Edema: limb (General disorders) | 13 | 21 | 12 | 0 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 203 | 191 | 36 | 5 | 7 | 1
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 24 | 35 | 10 | 1 | 3 | 1
Pain - Chest/thorax NOS (General disorders) | 17 | 15 | 7 | 0 | 1 | 0
Pain-Other (General disorders) | 24 | 29 | 7 | 0 | 1 | 0
Rigors/chills (General disorders) | 20 | 17 | 11 | 2 | 4 | 1
Syndromes-Other (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 5 | 6 | 4 | 0 | 0 | 0
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Eye NOS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 4 | 3 | 0 | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Skin (Infections and infestations) | 1 | 4 | 3 | 0 | 0 | 0
Infection with unknown ANC - Ureter (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Infection-Other (Infections and infestations) | 6 | 14 | 4 | 0 | 0 | 0
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 1 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 68 | 49 | 13 | 2 | 4 | 0
AST, SGOT (Investigations) | 55 | 41 | 9 | 2 | 4 | 0
Alkaline phosphatase (Investigations) | 38 | 14 | 7 | 2 | 3 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 3 | 4 | 2 | 1 | 0 | 0
CD4 count (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 0 | 7 | 0 | 0 | 1 | 0
Creatinine (Investigations) | 12 | 9 | 5 | 2 | 2 | 1
Leukocytes (total WBC) (Investigations) | 212 | 188 | 45 | 7 | 6 | 1
Lipase (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Lymphopenia (Investigations) | 80 | 94 | 32 | 4 | 6 | 1
Metabolic/Laboratory-Other (Investigations) | 11 | 7 | 5 | 0 | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 250 | 213 | 41 | 9 | 7 | 1
PTT (Partial thromboplastin time) (Investigations) | 3 | 1 | 3 | 0 | 0 | 0
Platelets (Investigations) | 19 | 23 | 44 | 2 | 3 | 1
Weight gain (Investigations) | 18 | 26 | 2 | 0 | 0 | 0
Weight loss (Investigations) | 11 | 12 | 1 | 1 | 1 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 36 | 35 | 13 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 42 | 47 | 13 | 3 | 3 | 0
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 30 | 32 | 16 | 2 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 10 | 5 | 1 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 69 | 82 | 23 | 4 | 5 | 0
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 | 9 | 5 | 2 | 1 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 | 2 | 4 | 0 | 1 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 | 5 | 5 | 1 | 1 | 0
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 | 7 | 5 | 0 | 0 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 12 | 19 | 22 | 1 | 3 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 19 | 18 | 10 | 1 | 2 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0 | 0
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4 | 7 | 6 | 2 | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 27 | 24 | 9 | 1 | 2 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 19 | 22 | 22 | 3 | 2 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 7 | 6 | 3 | 0 | 0 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 18 | 21 | 6 | 0 | 2 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 31 | 30 | 12 | 2 | 2 | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 39 | 45 | 9 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 30 | 25 | 12 | 2 | 1 | 0
Neuropathy: motor (Nervous system disorders) | 9 | 14 | 1 | 2 | 2 | 0
Neuropathy: sensory (Nervous system disorders) | 85 | 103 | 31 | 6 | 5 | 1
Ocular/Visual-Other (Nervous system disorders) | 10 | 15 | 2 | 0 | 0 | 1
Pain - Head/headache (Nervous system disorders) | 47 | 40 | 12 | 4 | 2 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 38 | 35 | 8 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 44 | 48 | 12 | 1 | 0 | 0
Libido (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Mood alteration - agitation (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0
Mood alteration - anxiety (Psychiatric disorders) | 21 | 25 | 8 | 1 | 1 | 0
Mood alteration - depression (Psychiatric disorders) | 11 | 14 | 5 | 0 | 1 | 0
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 1 | 0
Pain - Urethra (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 5 | 6 | 4 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12 | 24 | 3 | 0 | 1 | 1
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 72 | 13 | 0 | 3 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 56 | 70 | 17 | 1 | 2 | 0
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 0 | 0 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 4 | 0 | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 3 | 0 | 0 | 0
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 5 | 16 | 2 | 0 | 2 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 0 | 0 | 0
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 14 | 15 | 3 | 0 | 0 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 80 | 97 | 16 | 2 | 3 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 | 18 | 2 | 0 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 9 | 32 | 4 | 1 | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 21 | 20 | 2 | 2 | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 41 | 48 | 9 | 1 | 1 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 | 9 | 3 | 0 | 0 | 0
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 31 | 33 | 12 | 2 | 0 | 1
Hot flashes/flushes (Vascular disorders) | 7 | 17 | 7 | 1 | 1 | 0
Hypertension (Vascular disorders) | 4 | 6 | 2 | 1 | 2 | 0
Hypotension (Vascular disorders) | 6 | 5 | 2 | 1 | 1 | 0
Phlebitis (including superficial thrombosis) (Vascular disorders) | 5 | 9 | 2 | 1 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 6 | 8 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No